CLINICAL TRIAL: NCT00131209
Title: Lungwena Child Nutrition Intervention Study 3, LCNI-3. A Single-Centre Intervention Trial in Rural Malawi, Testing the Anthropometric and Health Benefits of Provision of Ready to - Use - Therapeutic Food RUTF as a Complementary Food
Brief Title: Trial to Test the Growth-Promoting Effect of Fortified Spreads When Used as Complementary Food for Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Academy of Finland (Other); Foundation for Paediatric Research, Finland (Other)
Responsible Party: Per Ashorn, University of Tampere Medical School, Finland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SA-1200720-3
Record Dates: First submitted 2005-08-16; First posted 2005-08-17 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-07

CONDITIONS: Malnutrition
Keywords: Infant; Sub-Saharan Africa; Complementary feeding; Malnutrition; Growth; Fortified spread; Haemoglobin
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: fortified spread (RUTF)
Dietary Supplement: maize and soy flour

SUMMARY:
This study tests the hypothesis that infants receiving fortified spread as a complementary food for one year grow better and do not become malnourished as often as infants who are provided with maize-soy flour for complementary porridge.

DETAILED DESCRIPTION:
Childhood undernutrition is very common in rural Malawi, like in many other countries in Sub-Saharan Africa. Usually, undernutrition develops between 6 and 24 months of age. By two years of age, 30-50% of all children in rural Malawi are undernourished, predisposing them to subsequent morbidity, developmental delay and mortality. Urgent interventions are needed but the magnitude of the problem precludes a hospital-based management strategy. Therefore, emphasis must be on prevention and early home-based rehabilitation of children with mild-to-moderate malnutrition. However, the options for community based approaches are not as developed as those for institutional management of undernutrition.

The present study tests a recently developed nutrient -dense spread, ready-to use- therapeutic food (RUTF), which offers a potential solution to home based nutrition rehabilitation. The concept has previously been shown to work not only in therapeutic feeding of undernourished children in nutrition rehabilitation units in Malawi but also home based supplementation of undernourished children in Mangochi District, southern Malawi. In the present study the investigators will test the efficacy in growth promotion and other health benefits of this product when provided as a complementary food to infants between 6 and 18 months of age.

The study will be conducted in Lungwena area, Mangochi District, rural Malawi. A total of 180 6-month old infants will be enrolled and randomised to three groups receiving different daily food supplements for 12 months. Children in group-one (control group) will receive 75g of maize/soy flour daily. Children in group-two will receive 25g RUTF daily and children in group-three will receive 50g RUTF daily for a period of 12 months. The food supplements will be delivered to the participant's home at weekly intervals.

All children will undergo medical and anthropometric examinations at 4-monthly intervals and disease symptoms monitoring every week. Dietary intake assessments will be conducted at 12 and 15 months of age. A random sample of 36 children will undergo breast milk intake assessments before the start of food supplementation and during food supplementation. A blood sample will be collected at the beginning and end of the study to measure blood haemoglobin and serum ferritin concentrations and test human immunodeficiency virus [HIV] (at 6 and 18 months).

The impact of the dietary interventions will be primarily assessed by comparing weight gain in the three intervention groups. Secondary outcomes include length gain, incidence of moderate underweight, stunting and wasting, cognitive and motor development at the end of trial and changes in blood haemoglobin and serum ferritin concentration. The study will also produce descriptive data on morbidity and intake of breast milk and other foods during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from at least one guardian
* Ages 5.50 months to 6.49 months
* Availability during the period of the study
* Permanent resident of the area

Exclusion Criteria:

* WHZ < -2.0 z-scores or presence of oedema
* History of peanut allergy
* Severe illness warranting hospital referral
* Concurrent participation of the child in another clinical trial with intervention to the child

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180
Dates: Start 2004-10; Primary Completion 2006-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Weight gain during the 12-month follow-up (in grams)

SECONDARY OUTCOMES:
Length gain during the study period (cm)
Cognitive and motor developmental score at the end of trial
Change in blood haemoglobin concentration during the study period (g/l)
Change in serum ferritin concentration during the study period (µg/l)
Mean change in anthropometric indices (weight-for-age z-score [WAZ], weight-for-height z-score [WHZ] and height-for-age z-score [HAZ])
Incidence of undernutrition, stunting and wasting (WAZ, WHZ or HAZ < -2.0)

CONTACTS AND LOCATIONS:
Overall Officials: Per Ashorn, MD, PhD, Study Director — University of Tampere, Medical School; Kenneth Maleta, MBBS, PhD, Principal Investigator — Kamuzu University of Health Sciences
Locations (1):
- College of Medicine, University of Malawi, Mangochi, Mangochi District, Malawi

REFERENCES:
- [Derived] Phuka JC, Maleta K, Thakwalakwa C, Cheung YB, Briend A, Manary MJ, Ashorn P. Postintervention growth of Malawian children who received 12-mo dietary complementation with a lipid-based nutrient supplement or maize-soy flour. Am J Clin Nutr. 2009 Jan;89(1):382-90. doi: 10.3945/ajcn.2008.26483. Epub 2008 Dec 3. PMID 19056572
- [Derived] Phuka JC, Maleta K, Thakwalakwa C, Cheung YB, Briend A, Manary MJ, Ashorn P. Complementary feeding with fortified spread and incidence of severe stunting in 6- to 18-month-old rural Malawians. Arch Pediatr Adolesc Med. 2008 Jul;162(7):619-26. doi: 10.1001/archpedi.162.7.619. PMID 18606932
- See also: College of Medicine home page — http://www.medcol.mw/